CLINICAL TRIAL: NCT02515331
Title: A Randomized, Sponsor Open, Site and Subject Double Blind, Parallel Group, Placebo-controlled Study to Evaluate the Safety and Efficacy of LHW090 After 4 Weeks Treatment in Patients With Resistant Hypertension
Brief Title: Safety and Efficacy Study of LHW090 in Resistant Hypertension Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLHW090X2202; 2015-001890-42 (EudraCT Number)
Record Dates: First submitted 2015-07-31; First posted 2015-08-04 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2018-06

CONDITIONS: Patients, Resistant Hypertension
Keywords: resistant hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LHW090 100 mg (Experimental): LHW090 100 mg once daily for 28 days
  Interventions: Drug: LHW090
- LHW090 200 mg (Experimental): LHW090 200 mg once daily for 28 days
  Interventions: Drug: LHW090
- Placebo (Placebo Comparator): Matching placebo to LHW090 oral dose for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LHW090 — Capsule - oral dose
  Arms: LHW090 100 mg; LHW090 200 mg
Drug: Placebo — Capsule - oral dose
  Arms: Placebo

SUMMARY:
The purpose of the present study was to determine whether LHW090 displays the clinical safety and efficacy profile to support further development in patients with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 40 to 85 years inclusive.
* • Patients with uncontrolled hypertension (here defined as having a mean daytime systolic BP ≥ 135 mmHg by ABPM at screening) despite treatment with a stable (at least 1 month) regimen that includes an optimal dose of an ARB plus a diuretic plus at least one additional class of anti-hypertensive medication.

For the purposes of this trial, optimal doses of anti-hypertensive medications are defined as:

* the highest dose listed in the clinical practice guideline from the American Society for Hypertension and the International Society for Hypertension or
* the highest allowable prescribed dose per the manufacturer's label or
* the highest dose tolerated by an individual patient or
* the highest dose appropriate for an individual patient in the judgment of the Investigator
* Subjects must weigh at least 45 kg to participate in the study and must have a body mass index (BMI) within the range of 18-38 kg/m^2.

Exclusion Criteria:

* Patients with an estimated GFR <60 ml/min/1.73m^2.
* Use of angiotensin converting enzyme inhibitors (ACE-inhibitors). Note: Patients who discontinue their ACE-inhibitor and substitute with an angiotensin receptor blocker may be eligible to be re-screened provided their anti-hypertensive regimen has been stable for at least 1 month. Any substitutions or changes to a patient's anti-hypertensive regimen should be done under the guidance of the patient's treating physician.
* Severe hypertension as defined by systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg at screening.
* A history of secondary hypertension of any etiology including but not limited to unilateral or bilateral renal artery stenosis, polycystic kidney disease, coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, pheochromocytoma, and drug-induced hypertension.
* Known current significant left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy or significant severe valvular disease on prior or current echocardiogram).
* A history of known moderate or malignant retinopathy defined as moderate (retinal signs of hemorrhage), microaneurysms, cotton-wool spots, hard exudates, or a combination thereof) or malignant (signs of moderate retinopathy plus swelling of the optic disk). Patients with a stable ophthalmologic history in the past 6 months are eligible.
* To facilitate ABPM assessment, an upper arm circumference greater than 42 cm.
* History within the previous 6 months of myocardial infarction, coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), hypertensive encephalopathy, stroke, or transient ischemic attack (TIA).

Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.

• Women of child-bearing potential

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (7):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, North Hollywood, California
  - Novartis Investigative Site, Atlantis, Florida
  - Novartis Investigative Site, Daytona Beach, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Knoxville, Tennessee
- Novartis Investigative Site, Gentofte Municipality, Denmark
- Novartis Investigative Site, Paris, France
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Homburg
- Novartis Investigative Site, Meibergdreef 9, Netherlands, Netherlands
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Lausanne

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=304

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1:2 ratio to LHW090 100 mg, LHW090 200 mg and placebo, respectively.
Period: Overall Study
Arm/Group | LHW090 100 mg | LHW090 200 mg | Placebo
Started | 17 | 15 | 32
Primary Pharmacodynamic Analysis Set | 15 | 14 | 29
Pharmacokinetic (PK) Analysis Set | 17 | 15 | 0
Completed | 15 | 15 | 28
Not Completed | 2 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 0 | 3
Not completed — Adverse Event | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LHW090 100 mg | LHW090 200 mg | Placebo | Total
Number analyzed (Participants) | 17 | 15 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (8.42) | 61.8 (5.16) | 64.4 (9.56) | 63.8 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13 | 26
  Male | 13 | 6 | 19 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 7 | 14 | 25
  White | 11 | 7 | 18 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reported Adverse Events (AEs), Serious Adverse Events (SAEs) and Deaths
Description: Number of participants with AEs, SAEs and deaths were assessed.
Time Frame: 6 months
Population: Safety analysis set: included all participants who were randomized.
Measure: Number; unit: Participants
Arm/Group | LHW090 100 mg | LHW090 200 mg | Placebo
Number analyzed (Participants) | 17 | 15 | 32
Participants
  AEs | 12 | 3 | 14
  SAEs | 0 | 0 | 0
  Deaths | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Mean Daytime Blood Pressure
Description: Change in the 12 hour average of systolic blood pressure (SBP) measured by ambulatory blood pressure was defined as the 12 hour daytime average SBP on Day 28 minus the 12 hour daytime average SBP on Day -1. monitoring (ABPM). A negative change from baseline indicates improvement.
Time Frame: Baseline, day 27
Population: The primary pharmacodynamics (PD) analysis set, which included patients that received study drug with any available PD data, was considered for the analysis. Only patients with values on both baseline and day 27 were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LHW090 100 mg | LHW090 200 mg | Placebo
Number analyzed (Participants) | 15 | 13 | 28
mmHg | -9.41 (8.379) | -16.84 (7.678) | -0.79 (10.555)
Statistical Analysis 1: Comparison: LHW090 100 mg vs Placebo; Test type: Superiority; p = 0.002, Longitudinal repeated measures mixed eff — 1-sided p-value; Mean Difference (Net) = -8.555, 95% CI 2-sided [-14.388 to -2.722], Standard Error of Mean 2.9077
Statistical Analysis 2: Comparison: LHW090 200 mg vs Placebo; Test type: Superiority; p < 0.001, Longitudinal repeated measures mixed eff — 1-sided p-value; Mean Difference (Net) = -14.727, 95% CI 2-sided [-20.852 to -8.602], Standard Error of Mean 3.0548

3. Secondary Outcome: Pharmacokinetics of LHW090/LHV527 in Plasma: Observe Maximum Plasma Concentration Following LHW090 at Steady State in Patients (Cmax)
Description: Blood samples were collected to assess Cmax.
Time Frame: Within 60 min prior to dosing, post dose: +/- 5 min up to 3 hrs, +/- 10 min from ≥3 hrs up to 12 hrs on Day 1 and Day 28
Population: The PK analysis set, which included participants with at least one valid PK concentration measurement and no major protocol deviations affecting PK data, was considered. Only participants with available PK data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LHW090 100 mg | LHW090 200 mg
Number analyzed (Participants) | 17 | 15
ng/mL
  LHW090, day 1: number analyzed (Participants) | 7 | 9
  LHW090, day 1 | 3620 (1220) | 6340 (3440)
  LHW090, day 28: number analyzed (Participants) | 14 | 11
  LHW090, day 28 | 4190 (1740) | 7340 (4300)
  LHV527, day 1: number analyzed (Participants) | 7 | 10
  LHV527, day 1 | 5040 (1770) | 6330 (3700)
  LHV527, day 28: number analyzed (Participants) | 15 | 11
  LHV527, day 28 | 5240 (1960) | 9870 (1810)

4. Secondary Outcome: Pharmacokinetics of LHW090/LHV527 in Plasma: Time to Reach the Maximum Concentration After Administration of LHW090 (Tmax)
Description: Blood samples were collected to assess Tmax.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | LHW090 100 mg | LHW090 200 mg
Number analyzed (Participants) | 17 | 15
hour
  LHW090, day 1: number analyzed (Participants) | 7 | 9
  LHW090, day 1 | 2.08 [1.00 to 7.95] | 3.00 [2.00 to 8.08]
  LHW090, day 28: number analyzed (Participants) | 14 | 11
  LHW090, day 28 | 2.00 [1.00 to 3.00] | 2.92 [0.383 to 8.08]
  LHV527, day 1: number analyzed (Participants) | 7 | 10
  LHV527, day 1 | 3.07 [2.08 to 8.03] | 4.08 [1.00 to 8.50]
  LHV527, day 28: number analyzed (Participants) | 15 | 11
  LHV527, day 28 | 3.92 [1.17 to 8.00] | 4.00 [2.38 to 8.08]

5. Secondary Outcome: Pharmacokinetics of LHW090/LHV527 in Plasma: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast)
Description: Blood samples were collected to assess AUClast.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hr*ng/mL
Arm/Group | LHW090 100 mg | LHW090 200 mg
Number analyzed (Participants) | 17 | 15
Hr*ng/mL
  LHW090, day 1: number analyzed (Participants) | 7 | 9
  LHW090, day 1 | 12300 (3870) | 24500 (16000)
  LHW090, day 28: number analyzed (Participants) | 14 | 11
  LHW090, day 28 | 13700 (4370) | 24400 (11400)
  LHV527, day 1: number analyzed (Participants) | 7 | 10
  LHV527, day 1 | 25300 (11800) | 28700 (17900)
  LHV527, day 28: number analyzed (Participants) | 15 | 11
  LHV527, day 28 | 27700 (11600) | 52300 (14400)

6. Secondary Outcome: Pharmacokinetics of LHW090/LHV527 in Plasma: Last Measurable Plasma Concentration (Clast)
Description: Blood samples were collected to assess Clast.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LHW090 100 mg | LHW090 200 mg
Number analyzed (Participants) | 17 | 15
ng/mL
  LHW090, day 1: number analyzed (Participants) | 7 | 9
  LHW090, day 1 | 404 (358) | 1710 (1600)
  LHW090, day 28: number analyzed (Participants) | 14 | 11
  LHW090, day 28 | 682 (752) | 1790 (1740)
  LHV527, day 1: number analyzed (Participants) | 7 | 10
  LHV527, day 1 | 3490 (1700) | 4670 (3050)
  LHV527, day 28: number analyzed (Participants) | 15 | 11
  LHV527, day 28 | 3430 (1340) | 7840 (3130)

7. Secondary Outcome: Pharmacokinetics of LHW090/LHV527 in Plasma:Tlast
Description: Blood samples were collected to assess Tlast.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | LHW090 100 mg | LHW090 200 mg
Number analyzed (Participants) | 17 | 15
hour
  LHW090, day 1: number analyzed (Participants) | 7 | 9
  LHW090, day 1 | 8.00 [7.07 to 8.08] | 8.00 [7.83 to 8.50]
  LHW090, day 28: number analyzed (Participants) | 14 | 11
  LHW090, day 28 | 8.00 [4.00 to 8.50] | 8.00 [7.83 to 8.50]
  LHV527, day 1: number analyzed (Participants) | 7 | 10
  LHV527, day 1 | 8.00 [7.07 to 8.08] | 8.00 [7.83 to 8.50]
  LHV527, day 28: number analyzed (Participants) | 15 | 11
  LHV527, day 28 | 8.00 [4.00 to 8.50] | 8.00 [7.38 to 8.08]

ADVERSE EVENTS:
Time Frame: up to 28 days
Groups:
- LHW090 100mg: LHW090 100 mg once daily for 28 days
- LHW090 200mg: LHW090 200 mg once daily for 28 days
Arm/Group | LHW090 100mg | LHW090 200mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15 | 0/32
Other Adverse Events (participants affected / at risk) | 12/17 | 3/15 | 14/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LHW090 100mg (N=17) | LHW090 200mg (N=15) | Placebo (N=32)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 0 | 3
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 1
Haematocrit increased (Investigations) | 1 | 0 | 0
Haemoglobin increased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 1
Urethral pain (Renal and urinary disorders) | 1 | 0 | 0
Breast discomfort (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT02515331/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT02515331/SAP_001.pdf